CLINICAL TRIAL: NCT02421796
Title: Malnutrition In Non-Celiac Wheat Sensitivity Patients
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM08
Record Dates: First submitted 2015-04-08; First posted 2015-04-21 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Non-Celiac Wheat Sensitivity
Keywords: n Non-Celiac Wheat Sensitivity; Malnutrition; Celiac disease; Irritable Bowel Syndrome
MeSH Terms: conditions — Malnutrition; Celiac Disease; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy specimens will be obtained from the bulb and the second duodenal portion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NCWS patients: Consecutive adult patients with an irritable bowel syndrome (IBS)-like clinical presentation, according to Rome II criteria, and a definitive diagnosis of NCWS.
- CD patients: Sex- and age-matched subjects with CD, diagnosed according to standard criteria during the same study period and enrolled as first control group.
- IBS patients: Sex- and age-matched subjects with IBS unrelated to NCWS or other food 'intolerance', diagnosed according to standard criteria during the same study period and enrolled as second control group.

SUMMARY:
Non-celiac gluten sensitivity (NCGS) or 'wheat sensitivity' (NCWS) is included in the spectrum of gluten-related disorders. No data are available on the prevalence of low bone mass density (BMD) in NCWS. Our study aims to evaluate the prevalence of malnutrition in NCWS patients and search for correlations with other clinical characteristics. This prospective observation study will include 90 NCWS patients with irritable bowel syndrome (IBS)-like symptoms, 90 IBS and 90 celiac controls. Patients will be recruited at the Internal Medicine and at the Gastroenterology Units of the University of Palermo. Elimination diet and double-blind placebo controlled (DBPC) wheat challenge proved the NCWS diagnosis. All subjects underwent nutritional parameters measurement, duodenal histology, Human Leucocyte Antigen (HLA) DQ typing and body mass index (BMI) evaluation.

DETAILED DESCRIPTION:
Celiac disease (CD) has been reported to increase the risk of malnutrition due to malabsorption. More recently, it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. That previous study also showed a percentage of NCWS patients had weight loss and anemia: whether these depended on the intestinal malabsorption or not remains unclear. As yet no data are available on the presence and prevalence of low bone mass density (BMD) in NCWS patients. The aims of the present study is 1) to investigate the prevalence of malnutrition in NCWS patient and 2) to search for a possible correlation with other clinical characteristics, in particular the body mass index (BMI), of NCWS patients.

ELIGIBILITY:
Inclusion Criteria:

To diagnose NCWS the recently proposed criteria will be adopted. All the patients will meet the following criteria:

* negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies;
* absence of intestinal villous atrophy;
* negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection);
* resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms;
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As the investigators previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges will be performed too.

Additional inclusion criteria will be:

* age >18 years; follow-up duration longer than six months after the initial diagnosis;
* at least two outpatient visits during the follow-up period.

Exclusion Criteria:

* positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa;
* self-exclusion of wheat from the diet and refusal to reintroduce it, before entering the study;
* other "organic" gastrointestinal disorders;
* nervous system disease and/or major psychiatric disorder;
* physical impairment limiting physical activity;
* menopause;
* steroid and sex steroid therapy, hormone replacement therapy or ovariectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include consecutive adult patients with irritable bowel syndrome (IBS)-like clinical presentation, according to Rome II criteria, and a definitive diagnosis of NCWS, referred at the Internal Medicine and at the Gastroenterology Units of the University Hospital of Palermo, between may 2015 and may 2017.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | At baseline and at 24 months
  The BMI [weight (kg) to the square of the height (m2)]. According to the World Health Organization, patients will be categorized as underweight (BMI <18.5), normal BMI 18.5 to 24.9, overweight BMI 25 to 29.9 and obese 30 to 39.9, and extreme obesity >40.

SECONDARY OUTCOMES:
Change in triceps skinfold thicknesses | At baseline and at 24 months
  Triceps skinfold measurement, using tricipital skinfold together with arm circumference, will be recorded as index of lean mass. The investigators will use the standard formula: AMC (Arm Muscle Circumference, mm) = UAC (Upper Arm Circumference, mm) - π (3.14) x TSF (Triceps Skinfold, mm).
Change in biometric impedance | At baseline and at 24 months
  Biometric impedance analysis will be performed to estimate total body water, extracellular water, fat-free mass and body cell mass.
Change in serum albumin | At baseline and at 24 months
  Serum albumin levels will be assayed (references values 3.4-5.4 g/dL).
Change in serum transferrin | At baseline and at 24 months
  Serum transferrin levels will be assayed (references values 200-360 mg/dL).
Change in total serum cholesterol | At baseline and at 24 months
  Total serum cholesterol levels will be assayed (references values <200 mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — Department of Internal Medicine, Giovanni Paolo II Hospital, Via Pompei, Sciacca, Italy
Locations (2):
- Italy (2):
  - Antonio Carroccio, Sciacca, Agrigento
  - Pasquale Mansueto, Palermo

REFERENCES:
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, Mansueto P, D'Alcamo A, Iacono G. Non-celiac wheat sensitivity as an allergic condition: personal experience and narrative review. Am J Gastroenterol. 2013 Dec;108(12):1845-52; quiz 1853. doi: 10.1038/ajg.2013.353. Epub 2013 Nov 5. PMID 24169272
- [Result] Carroccio A, Brusca I, Mansueto P, D'alcamo A, Barrale M, Soresi M, Seidita A, La Chiusa SM, Iacono G, Sprini D. A comparison between two different in vitro basophil activation tests for gluten- and cow's milk protein sensitivity in irritable bowel syndrome (IBS)-like patients. Clin Chem Lab Med. 2013 Jun;51(6):1257-63. doi: 10.1515/cclm-2012-0609. PMID 23183757
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366